CLINICAL TRIAL: NCT05871749
Title: Effects of Hepatic Fibrosis on Quantifying Hepatic Steatosis Using the Ultrasound Attenuation Imaging in Patients With Chronic Hepatitis B: a Prospective Study
Brief Title: Effects of Hepatic Fibrosis on Hepatic Steatosis Using the Ultrasound Attenuation Imaging in Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: So Yeon Kim (Other)
Collaborators: Canon Medical Systems, Korea (Unknown)
Responsible Party: Sponsor-Investigator, So Yeon Kim, Clinical Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AsanMC_2D-SWE_ATI_CHB
Record Dates: First submitted 2023-05-10; First posted 2023-05-23 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hepatic Steatosis; Hepatic Fibrosis; Chronic Hepatitis b
Keywords: Ultrasound Attenuation Imaging
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pathological degree of hepatic steatosis and fibrosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator aimed to prospectively study the effect of the hepatic fibrosis on quantifying hepatic steatosis using ultrasound attenuation imaging (ATI value) in patients with chronic hepatitis B.

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection has been reported to be associated with the prevalence of non-alcoholic fatty liver disease (NAFLD). Prior studies demonstrate that concurrent fatty liver increases risk of hepatocellular carcinoma among patients with chronic hepatitis B. Therefore, quantification of hepatic steatosis and fibrosis in chronic hepatitis B patient has important clinical significance in active surveillance.

Ultrasound imaging provides reliable noninvasive quantification of hepatic steatosis and fibrosis. Attenuation imaging (ATI) reflects hepatic steatosis and 2D-shear wave elastography reflects hepatic fibrosis.

The potential interaction between of the hepatic fibrosis and the hepatic steatosis in chronic hepatitis B is not fully understood. The investigator investigated the effect of the hepatic fibrosis on quantifying hepatic steatosis using ultrasound attenuation imaging (ATI value) in patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B patients
* Who is scheduled for pathological exam such as liver biopsy or surgery, that can quantify hepatic steatosis and hepatic fibrosis
* Who submitted informed consent

Exclusion Criteria:

* Who underwent liver transplantation or right hemihepatectomy
* Huge hepatic mass or numerous cysts in right hepatic lobe, who is not eligible for measuring ultrasound attenuation imaging and Fibroscan
* High bleeding risk patients

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients, who is schedule for pathological exam such as liver biopsy or liver surgery
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Attenuation Coefficient (AC) value at liver parenchyma | During procedure
  decibel(dB)/cm/megahertz(MHz)
Pathological hepatic steatosis | During procedure
  Non-alcoholic Steatohepatitis(NASH) Clinical Research Network scoring system as follows: S0, <5%; S1, 5%-33%; S2, 34%-66%; S3, ≥67%
Pathological hepatic fibrosis | During procedure
  Meta-analysis of histological data in viral hepatitis(METAVIR) scoring system as follows: F0, no fibrosis; F1, portal fibrosis without septa; F2, portal fibrosis with rare septa; F3, numerous septa without cirrhosis; and F4, cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Soyeon Kim, Professor, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul, Songpa-gu , 88, Olympic-ro 43-gil
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No